CLINICAL TRIAL: NCT00003341
Title: The Effects of Procrit (Epoetin Alfa) on Hemoglobin Symptom Distress and Quality of Life During Chemotherapy in Lymphoma Patients With Mild to Moderate Anemia A Multicenter Trial
Brief Title: Epoetin Alfa in Treating Anemia in Patients With Lymphoma, Chronic Lymphocytic Leukemia, or Multiple Myeloma and Anemia Caused By Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: 97-125; MSKCC-97125; ORTHO-PR-96-27-031; RPCI-DS-97-38; NCI-G98-1436
Record Dates: First submitted 1999-11-01; First posted 2003-04-25 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Anemia; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; Waldenström macroglobulinemia; stage II multiple myeloma; stage III multiple myeloma; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anemia; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Epoetin Alfa

INTERVENTIONS:
Biological: epoetin alfa
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs such as epoetin alfa may relieve anemia caused by chemotherapy. The best time for giving epoetin alfa during chemotherapy is not yet known.

PURPOSE: Randomized phase III trial to study the effectiveness of epoetin alfa in treating anemia in patients with lymphoma, chronic lymphocytic leukemia, or multiple myeloma who are receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the hematologic response and transfusion requirements of patients with malignant lymphoma, chronic lymphocytic leukemia, or multiple myeloma with chemotherapy related moderate anemia treated with epoetin alfa.
* Determine the effect of moderate anemia on quality of life of these patients treated with this regimen.
* Correlate changes in quality of life with changes in anemia associated with treatment with epoetin alfa in these patients.
* Determine the effect of changing quality of life on health care resource utilization among these patients treated with epoetin alfa.

OUTLINE: This is a randomized, open label, multicenter study.

Patients are evaluated for anemia during their prescribed chemotherapy regimens at either 3 or 4 week intervals beginning week 3 or 4. Patients with hemoglobin levels of 10.0-12.0 g/dL are randomized to 1 of 2 treatment arms. Patients with hemoglobin levels greater than 12.0 g/dL are not randomized until their hemoglobin levels decrease to 12.0 g/dL or below.

* Arm I: Patients immediately receive epoetin alfa subcutaneously each week.
* Arm II: Patients are observed for 6-8 weeks and then hemoglobin levels are reevaluated. Patients whose hemoglobin levels decrease below 9.0 g/dL receive epoetin alfa subcutaneously each week. Patients whose hemoglobin levels are at least 9.0 g/dL are observed for another 3-4 weeks and then hemoglobin levels are reevaluated.

Patients receive epoetin alfa treatment for up to 15 or 16 weeks.

Qualify of life questionnaires are completed every 3 or 4 weeks until week 30 or 32.

Patients are followed through week 36.

PROJECTED ACCRUAL: A total of 275 patients (at least 130 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma (NHL), chronic lymphocytic leukemia, or multiple myeloma

  * Low grade, intermediate grade, or high grade (diffuse large cell immunoblastic only) NHL OR
* Histologically confirmed Hodgkin's disease with prior chemotherapy
* Evaluable lesion
* Must be scheduled for at least 1 myelosuppressive cytotoxic regimen (experimental chemotherapy regimens allowed) for at least 4-6 months
* No anemia predominantly due to factors other than cancer or chemotherapy (i.e.,iron or folate deficiencies, hemolysis, or gastrointestinal bleeding) NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* Transferrin saturation at least 20%
* Ferritin at least 50 ng/mL OR
* Adequate iron stores in bone marrow
* If transferrin saturation is less than 20% or ferritin is less than 50 ng/mL, investigator may utilize bone marrow evaluation results to determine whether iron stores are adequate
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled hypertension

Other:

* HIV negative
* No active, unresolved infection
* No hypersensitivity to mammalian cell derived products
* Must be able to read and understand English at a 6th grade level consistent with comprehending the quality of life questionnaires
* No other malignancy within past 5 years, except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent epoetin alfa independent of protocol
* No concurrent interferons and interleukins (occasional short term use may be permitted on a case by case basis)
* No prior peripheral blood stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior total lymphoid, extensive abdominal, or inverted Y radiotherapy

Surgery:

* Not specified

Other:

* At least 30 days since prior nonchemotherapy experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Estimated)
Dates: Start 1997-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (18):
- United States (18):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Division of Oncology, Palo Alto, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas